CLINICAL TRIAL: NCT06994533
Title: Comparative Study on the Effect of New Reconstruction Methods and Traditional Reconstruction Methods on Bone Reconstruction After Chest Wall Tumor Resection
Brief Title: Comparative Study on Different Bone Reconstruction After Chest Wall Tumor Resection
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Principal Investigator, Wu Weiming, Thoracic Surgery, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 20250418
Record Dates: First submitted 2025-05-11; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Chest Wall Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- new methods on bone reconstruction after chest wall tumor resection (Experimental): Using noose fixation for thoracic bone reconstruction
  Interventions: Procedure: methods on bone reconstrucion after chest wall tumor resection
- traditional methods on bone reconstruction after chest wall tumor resection (Active Comparator): Using bridging method for thoracic bone reconstruction
  Interventions: Procedure: methods on bone reconstrucion after chest wall tumor resection

INTERVENTIONS:
Procedure: methods on bone reconstrucion after chest wall tumor resection — Selecting appropriate implants for chest wall bone reconstruction

SUMMARY:
Chest wall tumors are one of the important diseases in thoracic surgery, and surgery is still the main treatment for this disease in clinical practice. Surgery for chest wall tumors requires extensive resection. However, the extensive chest wall defect formed after extensive resection can lead to the destruction of the integrity and stability of the chest wall, thus requiring chest wall reconstruction. The reconstruction of the chest wall after resection has always been a difficult point in chest wall tumor surgery, and the reconstruction of the chest wall bone is a key point in chest wall reconstruction. The goals of successful chest wall bone reconstruction include restoring chest wall rigidity, minimizing chest wall deformities, maintaining lung mechanics, and protecting thoracic organs. At present, traditional reconstruction methods are based on simulating and restoring the anatomical structure of the thoracic spine. For certain special areas of chest wall defects (such as posterior rib and paraspinal tumors), it is difficult to perform residual fixation; At the same time, traditional reconstruction methods suffer from insufficient stability after reconstruction, such as loosening, detachment, displacement, and even fracture. Therefore, it is necessary to design new chest wall reconstruction methods to meet clinical needs.

DETAILED DESCRIPTION:
Chest wall tumors are one of the important diseases in thoracic surgery, and surgery is still the main treatment for this disease in clinical practice. Surgery for chest wall tumors requires the adoption of appropriate treatment plans based on the pathological results of the tumor, the location of tumor growth, the degree of local invasion of the tumor, and the presence of metastasis at the time of tumor detection. More importantly, surgical resection of primary malignant tumors of the chest wall should be carried out under careful planning, as most patients only have one chance of cure, and it becomes very difficult to undergo reoperation after tumor recurrence or surgical failure. Moreover, even if these patients undergo reoperation, their prognosis is also poor. To ensure the thoroughness of the surgery, it is usually necessary to perform an extensive resection of the chest wall tumor. However, the extensive chest wall defect formed after extensive resection can lead to the destruction of the integrity and stability of the chest wall, and if not handled properly, adverse consequences may occur. If chest wall softening, abnormal breathing, and acute respiratory failure occur early after surgery, it will affect the therapeutic effect of the surgery; In the late postoperative period, chest wall deformities, pulmonary hernias, chronic respiratory dysfunction, and even scoliosis may occur, affecting the quality of life. The reconstruction of the chest wall after resection has always been a difficult point in chest wall tumor surgery, and the reconstruction of the chest wall bone is a key point in chest wall reconstruction. The goals of successful chest wall bone reconstruction include restoring chest wall rigidity, minimizing chest wall deformities, maintaining lung mechanics, and protecting thoracic organs. In clinical treatment, it has been found that traditional reconstruction methods are unable to perform residual fixation for certain special areas of chest wall defects (such as posterior rib paravertebral tumors); There are also defects in the stability of the reconstructed implant, such as loosening, detachment, displacement, and even fracture. Therefore, it is necessary to design new chest wall reconstruction methods to meet clinical needs.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years old, male or female not limited
2. Anesthesia ASA score I-II
3. Malignant tumor of soft tissue in the chest
4. Malignant tumors of ribs, rib cartilage, and sternum
5. Tumors with uncertain or unknown properties of ribs, rib cartilage, and sternum
6. Giant benign tumors of ribs, rib cartilage, and sternum
7. The preoperative examination results indicate that the tumor has not undergone distant metastasis
8. Willing to participate in the research and sign the informed consent form

Exclusion Criteria:

1. Patients with distant metastasis detected during preoperative examination
2. Inoperable tumor
3. During the examination, it was discovered that the patient had another type of malignant tumor present
4. ECOG 4
5. Suffering from active or chronic fungal/bacterial/viral infections
6. History of allergy to anesthesia related drugs
7. Heart and lung dysfunction, liver and kidney dysfunction, inability to tolerate surgery
8. Patients with mental disorders who are unable to cooperate with treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Stability of implants | 3 years
  The occurrence of detachment, displacement, and fracture of implants during follow-up in patients undergoing chest wall tumor surgery after receiving a new reconstruction method

SECONDARY OUTCOMES:
Respiratory discomfort | 3 years
  Patient's respiratory discomfort in a calm state or walking state, measured as mild, moderate, or sereve after reconstruction surgery
Postoperative complications | 3 years
  Pulmonary infection, atelectasis, pleural effusion, respiratory failure, postoperative drainage tube removal time, length of hospital stay
Complications of implants | 3 years
  Fracture, displacement, infection, and compatibility of implants
Postoperative physical function status | 3 years
  Karnofsky scoring scale
Quality of life | 3 years
  EQ-5D-5L scoring scale, postoperative chronic pain level, postoperative recovery of daily work, postoperative changes in lung function (forced vital capacity FVC, first second forced vital capacity FEV1)
Postoperative chronic pain | 3 years
  NRS（Numberical rating scale）, postoperative recovery of daily work, postoperative changes in lung function (forced vital capacity FVC, first second forced vital capacity FEV1)
Postoperative recovery of daily work | 3 years
  The time from the day of surgery to the resumption of normal work, postoperative changes in lung function (forced vital capacity FVC, first second forced vital capacity FEV1)
Postoperative changes in lung function | 3 years
  FVC（forced vital capacity FVC） and FEV1（first second forced vital capacity）at 1 month, 3 months, 6 months, 1 year, 1.5 years, 2 years, and 3 years after surgery
chest wall discomfort in patients after reconstruction surgery | 3 years
  Patient chest wall discomfort in a calm or walking state, measured as mild, moderate, or severe after reconstrcution surgery
Chest wall appearance after reconstruction surgery | 3 years
  The degree of recovery of chest wall appearance after surgery is evaluated based on three criteria: satisfactory, moderately satisfactory, and unsatisfactory.

IPD SHARING:
Plan to Share IPD: No